CLINICAL TRIAL: NCT04413071
Title: Cardiac Involvement in Coronavirus (SARS-Cov-2) Infected Health Care Workers: The CCC Study
Brief Title: Cardiac COVID-19 Health Care Workers
Acronym: CCC
Status: Completed | Type: Observational
Sponsor: AORTICA Group (Other)
Collaborators: Salamanca University Hospital (Other); Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, Director of the Cardiology Department, Professor of Medicine, Salamanca University Hospital
Other Study IDs: CCC_2020
Record Dates: First submitted 2020-05-23; First posted 2020-06-02 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: SARS-CoV 2; COVID-19; Coronavirus; Cardiac Magnetic Resonance; Myocarditis; Cardiac Anomaly
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Myocarditis; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Analysis of immunity polymorphisms including low-resolution HLA typing and genotyping of KIR genes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health care workers: Health care workers from the University Hospital of Salamanca who have passed SARS-CoV-2 infection.
  Interventions: Other: Passed infection of SARS-CoV-2

INTERVENTIONS:
Other: Passed infection of SARS-CoV-2 — This is an observational design. Participants have passed infection from SARS-CoV-2 and a cardiac assessment is performed.

SUMMARY:
The study will analyze the prevalence of cardiac involvement of health care workers from the University Hospital of Salamanca (HUSA) who have overcome SARS-CoV-2 infection. Participants will undergo a clinical evaluation, electrocardiogram (EKG), cardiac magnetic resonance (CMR) and blood analysis including NT-proBNP, troponin, cellular and humoral immunity and genetics.

DETAILED DESCRIPTION:
Most people infected with SARS-CoV-2 experience mild, self-limiting symptoms that have been managed in an outpatient setting and therefore have not undergone routine cardiac evaluation with EKG or cardiac imaging test. Similarly, although the emphasis has been placed on evaluating patients with severe respiratory symptoms, most of these patients have also not undergone cardiac imaging tests and; therefore, in both scenarios, possible myocarditis has not routinely evaluated.

The present study is designed to characterize cardiac involvement in individuals who have overcome the SARS-CoV-2 infection.

For that aim, the study is designed as an observational cross-sectional study. The target population are HUSA healthcare workers who have overcome SARS-CoV-2 infection, either symptomatic or asymptomatic, either having required hospital admission or not. Participants will undergo a clinical evaluation, electrocardiogram (EKG), cardiac magnetic resonance (CMR) and blood analysis including NT-proBNP, troponin, cellular and humoral immunity and genetics.

Main objectives of the study are to address the prevalence of myocardial damage suggestive of myocarditis and to address the prevalence of pericarditis in HUSA health care workers; both related to the systemic immune response to SARS-CoV-2 infection. As secondary objectives the study will further address other cardiac affections including: rhythm or conduction disorders, ischemic heart disease, dilatation of the right chambers, valve disease and will analyze the relationship between humoral and cellular immunity and the presence of cardiac involvement, and the genetic susceptibility in the development of cardiac involvement after SARS-CoV-2 infection.

The study will recruit 141 participants: 47 symptomatic hospitalized health care workers, 47 asymptomatic non-hospitalized health care workers, 47 asymptomatic health care workers

ELIGIBILITY:
Inclusion Criteria:

* Have overcome the SARS-CoV-2 infection meeting any of the following criteria (i) positive result on a reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay of a specimen collected on a nasopharyngeal swab followed by a second negative RT-PCR and at least 14 days from this negative RT-PCR; (ii) presence of IgM antibodies and negative RT-PCR after the antibody assessment; (iii) presence of neutralizing IgG antibodies and absence of IgM.
* stable clinical situation, which allows performing a CMR.
* signature of informed consent.

Exclusion Criteria:

* Presence of IgM antibodies without negative subsequent RT-PCR.
* Contraindications to perform RMC: (i) gadolinium allergy, (ii) presence of metallic material in the body, such as plates, screws, incompatible pacemakers, etc. (iii) claustrophobia, (iv) severe kidney failure, (v) severe liver failure, (vi) sickle cell anemia

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are Salamanca´s healthcare workers who have overcome SARS-CoV-2 infection, either symptomatic or asymptomatic, either having required hospital admission or not.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Myocarditis | up to 3 months
  Prevalence of myocardial damage suggestive of myocarditis assessed by cardiac magnetic resonance
Pericarditis | up to 3 months
  Prevalence of pericarditis assessed by clinical criteria

SECONDARY OUTCOMES:
Atrial fibrillation | up to 3 months
  Prevalence of atrial fibrillation on EKG
Ischemic heart disease | up to 3 months
  Prevalence of ischemic heart disease assessed by cardiac magnetic resonance
Dilatation of right heart chambers | up to 3 months
  Prevalence of dilatation of right heart chambers assessed by cardiac magnetic resonance
Valvular hear disease | up to 3 months
  Prevalence of valvular heart disease assessed by cardiac magnetic resonance
Rhythm disorders | up to 3 months
  Prevalence of prolonged QT interval on EKG

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided